CLINICAL TRIAL: NCT01847937
Title: Magnetic Resonance Diagnostics of Diabetic Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Michael Vaeggemose, Research Assistant, Aarhus University Hospital
Other Study IDs: 1-10-72-85-13; VEK: 1-10-72-85-13 (Other Grant/Funding Number: UNIK Partnership)
Record Dates: First submitted 2013-04-12; First posted 2013-05-07 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Polyneuropathy; Hereditary Axonal Neuropathy; Hereditary Demyelinated Neuropathy; Polyneuropathy, Inflammatory Demyelinating, Chronic
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Neuropathies; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample less then 250ml to determine Hba1c (blood glucose level).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Diabetics Type I non-neuropathic: Diabetics with type 1 diabetes and without neuropathy
- Diabetics Type II non-neuropathic: Diabetics with type 2 diabetes without neuropathy
- Diabetics Type I neuropathic: Diabetics with type 1 diabetes and neuropathy
- Diabetics Type II neuropathic: Diabetics with type 2 diabetes and neuropathy
- Hereditary axonal neuropathic
- Hereditary demyelinated neuropathic: This will mainly be patients with Chronic inflammatory demyelinating polyneuropathy (CIDP).

SUMMARY:
This project aims to develop high field MR techniques to detect nerve lesions in diabetic patients. The MRI findings will be compared to results from conventional evaluations and nerve conduction studies to determine the validity as part of a clinical practice.

DETAILED DESCRIPTION:
Background

Diabetes mellitus is a very frequent disorder with an estimated prevalence of 275,000 patients in Denmark. Diabetic peripheral neuropathy (DPN) is a late complication which often remains undiagnosed, but may occur in up to 40% of diabetic patients. Advanced neuropathy may induce irreversible damages to the nervous tissue, and to avoid further damages, early diagnosis is important followed by optimal treatment of diabetes. DPN is a common complication due to long term diabetes in both type 1 and type 2.

Nerve conduction studies (NCS) is the gold standard method to diagnose DPN. However, the technique is time consuming and introduces discomfort to the patient and, furthermore, early nerve dysfunction may not be detected by NCS. Magnetic resonance imaging (MRI) (3 Tesla) of peripheral nerves is a new technique entitled Magnetic resonance neurography (MRN). In recent studies MRN has documented morphological changes in individual nerve fascicles. In T2-weighted images hyperintensity is present in proximal parts of nerves from neuropathic patients as compared to healthy nerves. This hyperintensity is believed to reflect early and more widespread lesions to the nerve fascicles that are not detected by NCS. This is pointing towards MRN to become an important tool in the management of patient with peripheral neuropathies.

Recent technical development such as diffusion weighted imaging (DWI) and diffusion tensor imaging (DTI) are currently being evaluated for imaging of the peripheral nerve system. DTI is expected to provide information about the physiology of the nerves and may reveal vascular congestion such as; blockade of axoplasmic flow, leading to abnormal proximal accumulation of endoneurial fluid; and distal Wallerian degeneration changes. Fiber tracking used on DTI is clinically implemented in some cases of stroke, tumours, neuropathy surgery, and functional brain MR imaging. Additionally, fiber tracking has been used on neuropathic patients with carpal tunnel syndrome, but has yet to be used in DPN as a measure of physiological function of the peripheral nerves.

Investigator, sponsor and trail setting Patients will be recruited at Department of Endocrinology and Internal Medicine from a cohort of more than 1000 well-characterized diabetic patients. The main investigator finished his masters as a biomedical engineer at the MR Centre at Aarhus University Hospital where he specialized in MR scanning techniques and has since been working with research combining diabetes, neuropathy, MR techniques and image processing. The studies will be conducted in collaboration between Siemens AG, Copenhagen, Department of Endocrinology and Internal Medicine, Department of Neurology, MR Centre at Aarhus University Hospital, Department of Endocrinology and Internal Medicine at Odense University Hospital and Department of Neuroradiology at Heidelberg University Hospital.

The main researchers on the project are as follows:

Main Investigator Michael Vaeggemose, MSc, Biomedical Engineering Department of Neurology, Aarhus University Hospital, Denmark

Supervisor Henning Andersen Professor, MD, PhD, Neurologist Department of Neurology, Aarhus University Hospital, Denmark

Supervisor Niels Ejskjaer Associate Professor, MD, PhD, Endocrinologist Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Denmark

Supervisor Knud Yderstraede Associate Professor, MD, PhD, Endocrinologist Department of Endocrinology, Odense University Hospital, Denmark

Supervisor Steffen Ringgaard Associate Professor, PhD, MR Physicist The MR Centre, Aarhus University Hospital, Denmark

Objective

This project aims to develop high field MR techniques to detect nerve lesions in diabetic patients. The MRI findings will be compared to results from conventional evaluations and nerve conduction studies to determine the validity as part of a clinical practice.

Methods

Blood sample

For the diagnosis of diabetes, HbA1c is used. This is the measure of how much glucose binding to hemoglobin in the blood. Diabetics have a higher blood sugar levels than healthy, there is definitely a threshold for diabetes that are at glucose values exceeding 64mmol/mol (8%). HbA1c is determined from a blood sample.

Clinical neurological test

Diabetics with and without neuropathy, hereditary axonal and demyelinated nerve injury patients examined with a clinical neurological test of sensibility, muscle power and reflexes. Examination of reflexes in the arms and legs performed with reflex hammer while the assessment of muscle strength is performed by trial participants to stretch and bend the arms and legs during resistance from the examiner. The subjects' sensibility of the soles is tested with a cotton swab and test participant shall so indicate on the touch can be felt. Furthermore the trial participants' vibration sensitivity of the soles is tested with a tuning fork. There is a possibly that the test of the muscles subsequently lead to slight muscle soreness, but otherwise there will be no significant risks, side effects or discomfort associated with the clinical neurological testing.

Neurophysiological studies

The neurophysiological studies include electroneurography (ENG) and Motor Unit Number Estimate (MUNE) and Motor Unit Number Index (MUNIX). The neurophysiological studies performed at the Clinical Neurophysiology Department, Aarhus University Hospital using EMG-equipped Keypoint (Medtronic, Skovlunde, Denmark).

Electroneurography (Nerve conduction study)

Nerve conduction studies are performed with the department's standardized methods and include:

1. Motor nerve conduction study and F-waves with surface electrodes on the ulnar peroneus, bilateral and tibial nerve, bilaterally.
2. Sensory nerve conduction study with surface electrodes of the sural nerve, bilaterally.

Nerve conduction velocities, amplitudes of the sensory and motor potential, distal motor latencies and minimum F-wave latencies are the parameters to be evaluated with nerve conduction studies.

MUNE Multipoint Stimulation & MUNIX

Motor Unit Number Estimate (MUNE) provides information on the number of functioning motor units in the studied muscle. The estimate is based on the ratio of the maximum Compound Muscle Action Potential (CMAP) and an average of that muscle on Surface Motor Unit Potentials (SMUP). In the current study used Multipoint Stimulation (MPS) for the stimulation of a nerve of one lower limb and a nerve in one upper limb per. participant. There is a one supramaximal nerve stimulation whereby the maximum CMAP determined with surface electrodes.

Then the nerve is stimulated, starting from 0 mA and increasing intensity to the first all-or-nothing SMUP observed. The intensity varied further until the measured SMUP not show variation (alternation.) process is carried out by moving the electrode a few millimetres along the nerve. This is done until a representative number SMUP is measured approx. 10 per. nerve.

Motor Unit Number Index (MUNIX) is also a MUNE technique. There will be conducted one supramaximal nerve stimulation with surface electrodes to obtain CMAP in the same nerve as used above. The next stage is electromyography (EMG) with the inclusion of surface interference pattern in voluntary contraction, typically by 10 different contractions between 10% and 90% of maximal contraction force.

The neurophysiological studies (ENG, MUNE, MUNIX) takes a total of 2 hours per trial participant and performed at the bonded small surface electrodes, respectively in hands or feet.

Muscle potential and nerve potential recorded through these surface electrodes for stimulation of the nerve with brief surges through the skin. This feels like a beating or pressing in the skin and may be associated with mild discomfort. Otherwise, the studies are not associated with any kind of risk or side effects.

MR Neurography (MRN)

MRN study will be conducted at Magnetrom Skyra 3 Tesla MR scanner (Siemens AG, Erlangen, Germany), which is set up to perform a MRN protocol with the following 5 sequences.

1. DIXON
2. Spectral adiabatic inversion recovery (SPAIR)
3. Short tau inversion recovery (STIR)
4. T2-weighted turbo spin echo (T2 TSE)
5. Diffusion weighted imaging (DWI)

Before the scan test, the subject must complete and comply with the rules of MRI safety. A description of the MRI scanning process, alarm ball, and a description of the noises the scanner produces is described to the subject. MRI methods for visualization of nerves does not use contrast agents, which is advantageous in the study of diabetes patients who may have reduced kidney function. The subject is placed supine on a bed with legs towards the scanner. To minimize motion artefacts a light fixation of the lower leg with foam pads is used. Around the foam pads and lower extremities is a 16-channel Peripheral Angio Array coil (Siemens AG, Erlangen, Germany) or multiple 18-channel Body Matrix coils (Siemens AG, Erlangen, Germany) located. To avoid hearing damage is a hearing protector placed on the subject's ear. If problems occur the test subject can at any time squeeze the alarm ball which is located in one hand, with a pressure on it and a direct contact with the investigator will be created and the patient can be moved out of the scanner. The scanning process is expected to take 2 hours with changing cloth, instruction and scanning. MRI scans are not associated with any kind of risk or side effects.

Quantitative sensory testing

Quantitative sensory testing (QST) is used to determine vibration threshold via a computerized sensory evaluation system (CASE IV WR Medical Electronics, Stillwater, MN, USA). This study investigated the trial participants' ability to perceive vibrations caused respectively the dominant index finger and the non-dominant foot big toe. In addition, temperature variation and pain perception in unity describes the neurological affliction stage and scope. The test is evaluated to exceeding patient specific thresholds for normal sensitivity or the extent of the patient's reduced or exaggerated sensitivity. The thermal test is an electrode applied to the skin. By adjusting the voltage of the electrode modified heat of the electrode with a linear increasing or decreasing the development of 40 degrees per second. Meanwhile the patient will be asked if he feel a temperature discomfort. QST is not associated with side effects, risks or discomfort.

Isokinetic dynamometry

The trail subjects' muscular strength is determined by isokinetic dynamometry. The test measures the maximum isokinetic strength of the shoulder flexor and extensor muscles of the dominant arm and the ankle flexor and extensor muscles in the non-dominant leg. Trials participant contract the muscles one at a time during a resistance and the study consists of a maximum of eight repetitions. This is done with a Biodex System 3 PRO dynamometer (Biodex Medical Systems Inc. NY, USA) and follows a standardized protocol. In very rare cases, muscle strain and tendinitis (less than 2 ‰) may occur, further risk, side effects or discomfort is not associated with the use of isokinetic dynamometry.

Statistical considerations

Comparison between matched groups will be performed using conventional statistic methods unpaired t-test or non-parametric tests such as Wilcoxon signed-rank test. In variation analyses of several groups ANOVA and ANCOVA will be used. A significant difference of p-values below 0.05 has to be determined, to determine the validity of the findings. Comparing the conventional methods to the MRI method from the binary outcome of being healthy or suffer from DPN, given an estimated sensitivity of 1 and a Specificity of 0.7, makes it possible to determine the required sample size. From a McNemar's test with a significant level of 5% a power calculation were performed giving a needed sample size of at least 50 subjects (healthy and diabetic with and without neuropathy). Inclusion of patients with axonal and demyelinated nerve lesions, to compare the resemblance of solely axonal and demyelinated damage to diabetic peripheral neuropathy, is in its current numbers not based on a statistical power calculation.

Volunteers

The trail consists of patients with type I and type II diabetes, with and without neuropathy. Patients will be recruited at the Department of Endocrinology, Noerrebrogade 44, Aarhus University Hospital. Patients with hereditary axonal and demyelinated neuropathy will be included at the Department of Neurology, Noerrebrogade 44, Aarhus University Hospital. Healthy subjects will be recruited through public media. In the 3 year course of the study it is expected to include 90 diabetics with and without neuropathy, 10 patients with hereditary axonal neuropathy and 10 patients with demyelinated neuropathy, as well as 35 healthy control subjects. This amounts to a total of 145 subjects.

Side effects, risk and disadvantages

The clinic neurological examinations test the subjects' reflexes, muscle strength and sensibility. The test of muscle strength can cause light muscle aches, but otherwise there will be no significant risks, side effects or disadvantages connected to the clinic neurological tests.

Vibration threshold is determined through a computer based sensory evaluation system (CASE IV, WE Medical Electronics, Stilwater, MN, USA) and is not connected to significant risks, side effects or disadvantages.

For examination of muscle strength the Biodex System 3 PRO dynamometer (Biodex Medical Systems Inc. NY, USA) is used. I very rare cases muscle strain and tendonitis (less than 2 ‰) I connection to the examination, otherwise there will be no significant risks, side effects or disadvantages connected to tests.

The neurophysiological examinations (ENG, MUNE, and MUNIX) are performed with surface electrodes with short bursts of electrical current through the skin. It feels like a beating or pressing under or in the skin and can be connected to discomfort. Besides this the tests are not connected to significant risks, side effects or disadvantages.

MR scans is not connected to any known risks and the patients ears will be protected with soundproofing earplugs or headphones to avoid the discomfort in relation to the high sound the scanner makes during the scans. The patients head will be placed outside the scanner, with the legs in the scanner, removing the risk of making the patient feel claustrophobic.

The blood test can be connected to slight discomfort and a small risk of developing accumulation of blood and infection at the needle injection site. If any sign of infection (rash, heating, tenderness, swelling) the subject must seek the investigator or the emergency room. Det combined blood loss in connection to the blood test will not exceed 250ml, which is a lot less than a blood donation includes.

The blood test is analysed and destroyed after. A bio bank will not be established in this project.

Since there's no significant side effects and risks in participating in the project it is considered that the project is scientific ethically justifiable.

Economic conditions

Expenses in connection to the project are covered by the involved departments. The researchers have no economic conflict of interest in the project. Transport expenses in connection to oral information and examination is refunded in regard to the guidelines used at the departments. In regard to national guidelines the subjects will be paid compensation for their partition in the project.

Publication of results

The results will be published in a recognized international paper in account to the Vancouver regulations regardless of the results are positive, negative or inconclusive.

Do the subjects wish information about the project results they can inform the investigator and he will send the information to the interested subjects.

National ethical committee review

The project is reported and approved by the Danish Data Protection Agency, Danish National Committee on Health Research Ethics (nr. 1-10-72-85-13) and the department legislations.

Volunteer recruitment

Subjects with peripheral nerve disease and non-neuropathic diabetic patients are recruited in the clinic at the Department of Neurology and Medical Department of Endocrinology, Aarhus University Hospital. Relevant potential subjects will be identified through their planned visit to Neurological clinic or Endocrinology clinic. Potential subjects (healthy controls, diabetics and patients with peripheral nerve disease) will receive written information about the research project with a request to contact the main investigator Michael Vaeggemose per letter, e-mail or telephone if they want further information about the research project. Healthy control subjects will be recruited by posting information material on public bulletin boards and in the local newspaper, indicating the main investigators phone number and e-mail address. Potential volunteers who want further information about the project would then subsequently receive the written participant information and National Ethics Committees information in regard to participating in a health science research project, and call for an information interview. The potential subject has the opportunity to bring a companion to the information interview and is informed of the right to stop participating in the project is he/she chooses to.

The information interview is conducted by PhD students, MSc biomedical engineer, Michael Vaeggemose who with in depth knowledge and close association to the studio has the necessary academic qualifications to do so. The conversation held in a conference room in undisturbed environment at Aarhus University Hospital, where the potential trial participant has the opportunity to bring a companion. Indicated during the interview that there is a request for participation in a biomedical research project and given an oral understandable presentation of the research project without using technical terms. During the interview, there will be enough time for the subject to listen to the oral information and ask questions. The conversation adapted beneficiary's individual requirements in terms of experience, maturity, age, etc.. The interview will be based on the written participant information and will include any foreseeable risks, side effects, complications and inconveniences associated with participation in the research project and that there may be unforeseen risks and impacts associated with participation in the research project. Furthermore, it is stated that information about health conditions, purely private matters and other confidential information may be disclosed to and processed by persons responsible for carrying out a statutory quality of the study. The subject is informed also about the right to decline knowledge of new essential health data in the project.

After information interview the potential trial participants has at least 1 week to think before signing the consent form. The subjects may at any time without consequences withdraw from the research project. It is desired to gain access to patient records, as evidenced by the written patient information. After the information interview the participant will be informed if, during the completion of the study, new data on the risks, complications and disadvantages in the trials has changed significantly in regard to the subject's safety. In the event that the study show crucial information about the subject's state of health it will be disclosed to the individual trial participant, unless they unequivocally expressed that this is not desired. The subjects will be informed of the results and of any consequences for the individual. There will be, upon completion of the project, a short easy to understand report in Danish summarizing the project's main results, as the individual trial participant may obtain by contacting the projects main investigator (Michael Vaeggemose). If the research project is interrupted the trial participants will be notified of the reason for this.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes, without neuropathy
* Clinical diagnosis of type 2 diabetes, without neuropathy
* Clinical diagnosis of type 1 diabetes, with neuropathy
* Clinical diagnosis of type 2 diabetes, with neuropathy
* Clinical diagnosis of hereditary axonal neuropathy
* Clinical diagnosis of hereditary demyelinised neuropathy
* Healthy controls who do not use prescription drugs and are of normal weight (BMI between 20 and 30).

Exclusion Criteria:

* The second cause of the neuropathy.
* Persons who are under 18.
* Inability to perform nerve conduction study or magnetic resonance imaging.
* Patients with liver disease, hypothyroidism, current or past alcohol abuse, rheumatological diseases and vasculitis.
* Silver Treatment, in diabetics with wounds.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the 3 year course of the study it is expected to include 90 diabetics with and without neuropathy, 10 patients with hereditary axonal neuropathy and 10 patients with demyelinated neuropathy, as well as 35 healthy control subjects. This amounts to a total of 145 subjects.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Increase in magnetic resonance signal intensity of segmented nerves | within the first 20 days (plus or minus 6 days) after initial MR scan
  Magnetic resonance neurography signal intensities from the sciatic, peroneal, and sural nerve is increased in diabetic patients with peripheral neuropathy compared to healthy control subjects.

SECONDARY OUTCOMES:
Determine diffusion weighted magnetic resonance values according to neuropathy | within the first 20 days (plus or minus 6 days) after initial MR scan
  Diffusion weighted MR provides valuable physiological neuropathy information.
Examination of magnetic resoance morphological differences according to neuropathy | within the first 20 days (plus or minus 6 days) after initial MR scan
  Magnetic resonance neurography reveal significant variation in nerve lesions of patients with axonal, demyelinated, and diabetic peripheral neuropathy.
Correlation of magnetic resoance signal intensity value and nerve conduction thresholds | within the first 20 days (plus or minus 6 days) after initial MR scan
  The number of damaged nerve fascicles in the sciatic, peroneal, and sural nerve at diabetic patients examined with magnetic resonance images correlates with diabetic peripheral neuropathy examined with conventional tests, nerve conduction velocity, and quantitative sensory testing.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaeggemose, MSc, Principal Investigator — Department of Neurology, Aarhus University Hospital
Locations (5):
- Denmark (4):
  - Department of Endocrinology and Internal Medicine, Aarhus, Aarhus
  - Department of Neurology, Aarhus, Aarhus
  - Department of Neurophysiology, Aarhus, Aarhus
  - MR Centre, Aarhus, Aarhus
- Neurologische Universitätsklinik Heidelberg Abteilung für Neuroradiologie, Heidelberg, Baden-Wurttemberg, Germany